CLINICAL TRIAL: NCT04666961
Title: Impact of Neoadjuvant Hormonal Therapy on the Surgical Management of Extensive Ductal Carcinomas in Situ
Acronym: HORNEO01
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICO-2020-06
Record Dates: First submitted 2020-12-02; First posted 2020-12-14 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Ductal Carcinoma in Situ; Extensive Disease; Mastectomy
Keywords: Neoadjuvant hormonotherapy; Tamoxifen; Anastrozole; conservative surgery; Breast cancer; extensive microcalcifications
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Breast Neoplasms | interventions — Tamoxifen; Anastrozole

STUDY DESIGN:
Intervention Model Description: Patients with extensive ductal carcinoma in situ with an indication for mastectomy receiving neoadjuvant hormone therapy with Tamoxifen (non-menopausal patients) or Anastrozole (postmenopausal patients)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Extended ductal carcinoma in situ with mastectomy indication (Experimental): Patients receive 6 months of tamoxifen or anastrozole in a neoadjuvant situation.
  Tamoxifen and Anastrozole will be delivered in their original packaging at J0 and M3 :
  * Tamoxifen: box of tablets dosed at 20 mg
  * Anastrozole: box of tablets 1 mg. Tamoxifen will be initiated in premenopausal patients orally at a standard dose of 20mg/day as a single dose for 6 months.
  Anastrozole will be administered orally to postmenopausal patients at the standard dose of 1mg/day in a single dose for 6 months.
  Interventions: Drug: Tamoxifen 20 mg; Drug: Anastrozole 1Mg Tab

INTERVENTIONS:
Drug: Tamoxifen 20 mg — Tamoxifen will be initiated in non menopausal patients orally for 6 months in a neoadjuvant situation.
Drug: Anastrozole 1Mg Tab — Anastrozole will be initiated in menopausal patients orally for 6 months in a neoadjuvant situation.

SUMMARY:
Ductal carcinoma in situ (DCIS) accounts for approximately 20% of newly diagnosed breast cancer cases. Of these women, 20% require radical management in the form of mastectomy because of the extent of the lesions, which most often manifest as diffuse microcalcifications.

This mutilating surgical management contrasts with the excellent prognosis of this pathology and considerably alters the quality of life of patients.

Neoadjuvant hormone therapy has shown its efficacy in hormone-dependent infiltrating ductal carcinomas and offers the possibility of conservative surgery after hormone therapy.

Adjuvant hormone therapy with Tamoxifen or anti-aromatase drugs has shown its efficacy in the prevention of homo or contralateral recurrence.

The HORNEO 01 trial fits perfectly in the current context of surgical de-escalation of ductal carcinomas in situ. The objective of the study is to evaluate the impact of neoadjuvant hormone therapy on the surgical management of extensive DCIS.

DETAILED DESCRIPTION:
Description of the modalities for recruiting :

Following screening and discovery of a DCIS, patients are referred to the center for surgical management.

During a standard consultation, the surgeon presents the study to the patient who has been diagnosed with extensive DCIS with an indication for mastectomy. The surgeon provides the patient with the information note and the consent form to participate in the study. Once the consent form is signed by the patient and the investigator, the investigator prescribes a screening test to be performed within 30 days prior to the start of hormone therapy.

Screening assessment includes :

A clinical exam and a breast imaging exam (mammography and breast and axillary ultrasound). In case of a suspicious breast ultrasound image, microbiopsy will be performed to eliminate an infiltrating component.

One or more macrobiopsy. Each biopsied site will be located using an X-ray clip inserted at the time of sample.

A MRI post-macrobiopsy. Research of estrogen receptor expression

Once the investigator has verified and validated all the eligibility criteria, the patient will be included.

Prescriptions for Tamoxifen (non-menopausal patients) or Anastrozole (menopausal patients) are given to patients and dispensed by the center's pharmacy.

Monitoring during treatment :

Patients will benefit from imaging monitoring (Mammography, +/- breast ultrasound, +/- axillary ultrasound, MRI) at 3 months and 6 months during hormonotherapy.

In case of progression observed during treatment, hormone therapy will be stopped and you will then benefit from a mastectomy.

Surgery :

Mastectomy or tumorectomy will be performed according to the tumor response to hormone therapy observed on MRI.

All patients will benefit sentinel node detection. An additional axillary dissection will be performed based on the results of the sentinel node analysis.

Analysis of biomarkers and tumor microenvironment before and after treatment on diagnostic macrobiopsies and on tumorectomy or mastectomy will be performed at Institut de Cancérologie de l'Ouest.

Patients will be seen in postoperative consultation. Adjuvant treatments or re-surgical interventions will be prescribed, carried out, and the patients will be followed up and examined at 6 months after surgery or at the end of adjuvant treatments and then annually for 10 years (with control mammography).

Patients who have had conservative surgery will have an MRI at 6 months from the end of radiotherapy.

All patients will be asked to complete quality of life questionnaires at baseline, 6 and 12 months post-surgery, and annually for 9 years:

EORTC QLQ-C30 (up to 5 years only), Short Form (36) Health Survey questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Patient ≥ 40 years old
2. Histological diagnosis of ductal carcinoma in situ without infiltrating contingent
3. Clinical T0N0
4. Estrogen receptor positive (OR+) regardless of progesterone receptor (PR) status
5. Indication for mastectomy
6. DCIS visible on MRI performed with clip sequence
7. Effective contraceptive method for women of childbearing age who are sexually active and who have reported sexual activity.
8. Informing the patient and obtaining free, informed and written consent signed by the patient and the investigator.
9. Affiliated patient or beneficiary of the social security system.

Exclusion Criteria:

1. Invasive breast carcinoma
2. Lobular carcinoma in situ
3. pN+ patient
4. Indication for conservative surgery
5. Contraindications to anastrozole or tamoxifen
6. Concomitant treatments that may interact and reduce the efficacy of tamoxifen by interaction with cytochrome CYP2D6.
7. Histologically proven multifocal lesion
8. Contraindication to breast MRI (pace maker, heart valve, metallic implant, neuronal or peripheral stimulator, severe claustrophobia, ...)
9. History of homolateral breast cancer
10. Ongoing contralateral breast cancer
11. Known mutation BRCA1 BRCA2
12. Other cancer in progress at inclusion
13. Pregnant woman, or breastfeeding,
14. Persons deprived of liberty or under guardianship or trusteeship,
15. Impossibility to undergo the medical follow-up of the trial for geographical, social, psychic or psychiatric reasons.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Estimated)
Dates: Start 2021-02-03 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2033-08-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of neoadjuvant hormonotherapy | 6 months of hormonotherapy
  % of conservative surgeries performed after hormonotherapy

SECONDARY OUTCOMES:
Disease-free survival (DFS) | 5 and 10 years post-surgery
  DFS rates at 5 and 10 years post-surgery
Overall survival (OS) | 5 and 10 years post-surgery
  Survival rates at 5 and 10 years post-surgery
Pathologic Complete Response (pCR) | 6 months of hormonotherapy
  Pathologic complete response is defined as no residual invasive cancer in the surgical specimen
Predictive factors of response | 3 and 6 months of hormonotherapy
  Response is defined by the variation in the diameter of the longest dimension of the target lesion measured by MRI
Quality of Life (Qol) | At baseline, at 6 months and 12 months post-surgery, and then each year for 4 years
  EORTC QLQ-C30 questionnaire
Quality of Life (Qol) | At baseline, at 6 months and 12 months post-surgery, and then each year for 9 years
  SF-36 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Victoire BRILLAUD-MEFLAH, MD, Principal Investigator — Institut de Cancérologie de l'Ouest
Locations (8):
- France (8):
  - ICO - Site Paul Papin, Angers
  - Institut Bergonie, Bordeaux
  - Institut de cancérologie de Montpellier, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Institut Curie - Site de Paris, Paris
  - Hopital Saint Joseph, Paris
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - IUCT-O, Toulouse